CLINICAL TRIAL: NCT06693518
Title: A PHASE 1, OPEN-LABEL, RANDOMIZED, 2-PERIOD, 2-SEQUENCE, CROSSOVER STUDY TO ESTIMATE THE EFFECT OF IBUZATRELVIR ON THE PHARMACOKINETICS OF DABIGATRAN IN HEALTHY ADULT PARTICIPANTS
Brief Title: A Study to Learn About if the Study Medicine Called Ibuzatrelvir Changes How the Body Process the Other Medicine Dabigatran Etexilate in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: C5091010; 2024-517797-14-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2024-11-05; First posted 2024-11-18 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: SARS-CoV-2 Infections
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment A= Dabigatran Etexilate 150 mg (Experimental): Treatment A= Dabigatran Etexilate 150 mg
  Interventions: Drug: Treatment A
- Treatment B=Ibuzatrelvir 600 mg + Dabigatran Etexilate 150 mg (Experimental): Treatment B=Ibuzatrelvir 600 mg + Dabigatran Etexilate 150 mg
  Interventions: Drug: Treatment B

INTERVENTIONS:
Drug: Treatment B — Ibuzatrelvir 600 mg + Dabigatran Etexilate 150 mg
  Arms: Treatment B=Ibuzatrelvir 600 mg + Dabigatran Etexilate 150 mg
Drug: Treatment A — Dabigatran Etexilate 150 mg
  Arms: Treatment A= Dabigatran Etexilate 150 mg

SUMMARY:
This is a Phase 1, open-label, randomized, 2-period, 2-sequence, cross-over study to estimate the effect of ibuzatrelvir on the PK of dabigatran, a P-gp substrate, in healthy adult participants. Participants who discontinue from the study for non-safety reasons may be replaced at the Sponsor's discretion in collaboration with the investigator.

Healthy participants will be screened to determine eligibility within 28 days prior to study treatment. Participants will report to the CRU on Period 1 Day -1 in Period 1 and will be required to stay at the CRU until discharge Day 3 in Period 2.

This study will consist of two treatments. Treatment A: 150 mg of dabigatran etexilate; Treatment B: ibuzatrelvir 600 mg + 150 mg of dabigatran etexilate. The participants will be fasted overnight for at least 10 hours before administration of study intervention. Serial dabigatran samples will be collected up to 48 hours post-dose in both Period 1 and Period 2. Dosing of dabigatran in Period 1 and 2 will be separated by approximately 72h.

A follow-up (which may be a phone call) will be made to participants approximately 28 to 35 days from administration of the final dose of study intervention.

Approximately 20 participants will be enrolled in the study. PK samples will be collected for Dabigatran and Ibuzatrelvir as per SOA.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants 18 to 75 years of age, inclusive, at screening who are overtly healthy as determined by medical evaluation, including medical history, physical examination, laboratory tests, and standard 12-lead ECGs.
2. BMI of 17.5 to 32 kg/m2; and a total body weight >50 kg (110 lb).
3. Capable of giving signed informed consent.
4. Willing and able to comply with all scheduled visits, treatment plans, laboratory tests, lifestyle considerations, and other study procedures.

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing) and, in the judgment of the investigator, would make the participant inappropriate for entry into this study. Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy). History of HIV infection, hepatitis B, or hepatitis C. Positive testing for HIV, HBsAg, or HCVAb. Hepatitis B vaccination is allowed.
2. Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality or other conditions that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
3. Use of prescription or nonprescription drugs and dietary and herbal supplements within 28 days or 5 half-lives (whichever is longer) prior to the first dose of study intervention.
4. Participation in other studies involving study intervention within 30 days or 5 half-lives (whichever is longer) prior to study entry. Previous administration with an investigational product (drug or vaccine) within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer). Participation in studies of other investigational products (drug or vaccine) at any time during participation in this study.
5. Active bleeding or risk of bleeding, including prior personal or family history of abnormal bleeding, hereditary or acquired coagulation or platelet disorder or abnormal coagulation test (PT/INR or PTT/aPTT) greater than the upper limit of normal result at screening. Any significant risk factor for major bleeding, which may include but is not limited to current or recent GI ulceration, presence of malignant neoplasms at high risk of bleeding, recent brain or spinal injury, recent brain, spinal, or ophthalmic surgery, recent intracranial hemorrhage, known or suspected esophageal varices, arteriovenous malformations, vascular aneurysms, or major intraspinal or intracerebral vascular abnormalities.
6. A positive urine drug test. A single repeat for positive drug screen may be allowed.
7. Pregnant or breastfeeding women or evidence of positive pregnancy test at screening or Study Day -1.
8. Screening supine BP ≥ 140 mmHg (systolic) or ≥90 mmHg (diastolic) for participants <60 years and ≥150/90 mmHg for participants ≥60 years old, following at least 5 minutes of supine rest. If systolic BP is ≥ 140 or 150 mmHg (based on age) or diastolic BP is ≥ 90 mmHg, the BP should be repeated two more times, and the average of the three BP values should be used to determine the participant's eligibility.
9. An eGFR of <75 mL/min as determined by CKD-EPI equation using Screat as described in Section
10. Screening supine standard 12-lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, QTcF > 450 msec or QRS interval > 120 msec, complete LBBB, signs of an acute or indeterminate age myocardial infarction, ST-T interval changes suggestive of myocardial ischemia, second- or third-degree AV block, or serious bradyarrhythmias or tachyarrhythmias). If the uncorrected QT interval is > 450 msec, this interval should be rate-corrected using the Fridericia method only, and the resulting QTcF should be used for decision making and reporting. If QTcF exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated twice, and the average of the three QTcF or QRS values should be used to determine the participant's eligibility. Computer-interpreted ECGs should be overread by a physician experienced in reading ECGs before excluding a participant.
11. Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study-specific laboratory and confirmed by a single repeat test, if deemed necessary:

    AST or ALT ≥1.5 × ULN Total bilirubin ≥1.5 × ULN; participants with a history of Gilbert's syndrome may have a direct bilirubin measured and would be eligible for this study provided the direct bilirubin is ≤ ULN PT/INR or PTT/aPTT >1.0 × ULN
12. Participants who have recently underwent a surgery or invasive procedure prior to study enrollment, or who anticipate requiring it during study conduct, are ineligible for this study.
13. History of sensitivity reactions to dabigatran etexilate or any of the formulation components of ibuzatrelvir or dabigatran etexilate.
14. Have any medical conditions, medical history, or are taking any medications that are contraindicated in the dabigatran etexilate prescribing information.
15. History of alcohol abuse or repeated binge drinking and/or any other illicit drug use or dependence within 6 months of screening. Binge drinking is defined as a pattern of 5 (male) and 4 (female) or more alcoholic drinks in about 2 hours. As a general rule, alcohol intake should not exceed 14 units per week (1 unit = 8 ounces (240 mL) beer, 1 ounce (30 mL) of 40% spirit, or 3 ounces (90 mL) of wine).
16. Use of tobacco or nicotine-containing products in excess of the equivalent of 5 cigarettes per day or two chews of tobacco per day.
17. Investigator site staff directly involved in the conduct of the study and their family members, site staff otherwise supervised by the investigator, and sponsor and sponsor delegate employees directly involved in the conduct of the study and their family members.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-11-22 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Cmax | 0 - 48 hours
  Plasma Cmax (Maximum observed concentration) of Dabigatran with ibuzatrelvir (Test) versus without ibuzatrelvir (Reference)
AUCinf | 0 - 48 hours
  Plasma AUCinf of Dabigatran with ibuzatrelvir (Test) versus without ibuzatrelvir (Reference)

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | Day 1 till follow up visit (Day 28-35)
Incidence of clinical laboratory abnormalities | Day 1 till follow up visit (Day 28-35)
Incidence of vital sign abnormalities | Day 1 till follow up visit (Day 28-35)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - Brussels, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5091010